CLINICAL TRIAL: NCT05508230
Title: Clinical Study to Evaluate the Safety of the Investigational Product NASAL SPRAY Through of Assessments of Cutaneous Acceptability and Perceived Efficacy Under Normal Conditions of Use
Brief Title: Evaluation of Cutaneous Acceptability and Perceived Effectiveness of a Nasal Spray (Health Care Products)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herbarium Laboratorio Botanico Ltda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HB2053-23
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Acceptance, Social; Sensitivity, Contact
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Hyaluronic Nasal Spray

INTERVENTIONS:
Other: Hyaluronic Nasal Spray — Health care product - nasal application

SUMMARY:
This is a clinical study for health care product safety assessment. The research is going to conducted with 45 subjects, aged 18 to 70 years, women users of the product category, regardless of color/race, ethnicity, sexual orientation, classes and social groups and who must present all the other characteristics of the inclusion criteria and no exclusion characteristics. The product is applied under real conditions of use, in a panel of survey participants corresponding to the target consumers. Medical evaluation will be available throughout the study to assess possible adverse events. The main of the study is to observe the effects of the application of the product on the skin and prove the absence of irritability and/or allergy and perceived acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Phototype (Fitzpatrick): I to VI.
* User of the same product category.
* Have intact skin in the study region.
* Agree to adhere to the study procedures and requirements: study time, returns (after 28 days) to the laboratory to perform the study procedures, home use of the investigational product, filling in the use diary, not changing facial cosmetic habits during the period of study.
* Agree not to perform facial aesthetic dermatological treatments until the end of the study (28 days), such as: peelings, laser, fillers, use of any facial cosmetics.
* Agree to adhere to the requirements of the study in the fight against the COVID-19 pandemic, through preventive measures: use a mask according to WHO guidelines; use the mask while traveling to the research center and during the study procedures; maintain social distancing; wash hands frequently with soap and/or alcohol gel and go to the research center only at scheduled times to avoid agglomerations.
* Signing of the Free and Informed Consent Term (FICT).

Exclusion Criteria:

* Pregnant or lactating women.
* Skin tags in the experimental area that interfere in the assessment of possible skin reactions (pigmentation disorders, vascular malformations, scars, increased hairiness, large amounts of freckles and warts, sunburn).
* Presence of active dermatoses or skin lesions (local and/or disseminated) in the study region.
* Carriers of corneal ulcerations, keratoconus, blepharitis, meibomitis, pterygium, chemosis, hyperemia or other active eye diseases of moderate or severe intensity.
* History of ineffectiveness, allergic reactions, irritation or intense discomfort sensation to topical products: cosmetics or medicines.
* Expected vaccination during the study or up to 3 weeks before the study;
* History of pathologies aggravated or triggered by ultraviolet radiation.
* Use of non-steroidal anti-inflammatory drugs, corticosteroids, antihistamines, photosensitizers or immunosuppressants up to 2 weeks before the study.
* Facial aesthetic or dermatological treatment up to 4 weeks before the study.
* Hormonal treatments not stable in the last 3 months.
* Hyperpigmentation associated with the use of drugs such as tetracycline, phenothiazides, or amiodarone.
* Hyperpigmentation associated with photosensitivity.
* Actinic lichen planus;
* People directly involved in carrying out this study and their families.
* Be participating in another study.
* History of non-adherence or unwillingness to adhere to the study protocol.
* Intense sun exposure or tanning session up to 15 days before the initial assessment;
* Any condition not mentioned above that, in the opinion of the investigator, could compromise the evaluation of the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Erythema degree or absence | 28 days
  Erythema evaluation according to International Contact Dermatitis Research Group

CONTACTS AND LOCATIONS:
Locations (1):
- Kosmoscience Ciência e Tecnologia Cosmética Ltda, Campinas, São Paulo, Brazil